CLINICAL TRIAL: NCT03287739
Title: Recovery of Impairments Early After Stroke
Acronym: aRISE
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00889
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: Upper Extremity; Cohort Studies; Prognosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group study: Assessment of behavioral biometric impairments
  Interventions: Behavioral: Assessment of behavioral biometric impairments

INTERVENTIONS:
Behavioral: Assessment of behavioral biometric impairments — Assessment of behavioral biometric impairments

SUMMARY:
Upper limb recovery after stroke is highly predictable early after stroke. Nijland et al. showed that based on two simple clinical bedside tests - 'Shoulder Abduction' and 'Finger Extension' (the so called 'SAFE model' [Stinear et al., 2012]) - measured within the first 72 hours after stroke, ~87% of the patients could be correctly classified as either regaining or not regaining some dexterity (recoverers or nonrecoverers, respectively) (Nijland et al., 2010). This kind of information regarding the patients' functional prognosis allows proper discharge planning, setting realistic rehabilitation goals, and adequate patient information. However, the length of hospital stay after stroke has been decreasing. Therefore, knowledge is needed regarding the ability to make an accurate first prediction within the first 24 hours after stroke onset while using simple clinical bedside assessments. This would facilitate an earlier triage and with that, an accelerated and smooth transition of patients within the stroke care continuum. In addition, a first prediction within 24 hours poststroke has the potential to decrease health care expenses, as length of hospital stay after an acute stroke is ~30% of the total costs (i.e., direct and indirect costs) associated with stroke (Roger et al., 2012; Fattore et al., 2012).

The primary objective of aRISE is to determine the ability of the behavioral biometric impairments 'Shoulder Abduction' and 'Finger Extension' measured <24 hours poststroke to predict outcome of upper limb capacity 3 months after stroke. The secondary aim is to investigate the the added value of other simple clinical bedside tests for predicting outcome of upper limb capacity 3 months poststroke.

aRISE is a prospective longitudinal observational cohort study of 40 first-ever ischemic stroke patients, who will be assessed <24 hours, 7 days and 3 months after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* First-ever unilateral ischemic stroke in the middle cerebral artery territory <48 hours, confirmed by MRI-DWI and/or CT
* Age 18 years or older
* Able to follow one-staged commands
* NIHSS arm score ≥1
* Informed consent after participants' information

Exclusion Criteria:

* Modified Rankin Scale score >2 before stroke
* Neurological or other diseases affecting the upper limb(s) before stroke
* Intravenous line in the upper limb(s) which limits assessment
* Contra-indications on ethical grounds
* Expected or known non-compliance to participate in the observational study, severe drug or/and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-ever unilateral ischemic stroke patients, admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | 3 months poststroke
  Upper limb capacity
Fugl-Meyer Assessment | 3 months poststroke
  Upper limb motor function
Motricity Index | 3 months poststroke
  Upper limb motor function

OTHER OUTCOMES:
Surface Electromyography | 48 hours, 7 days, and 3 months poststroke
  Forearm skeletal muscle electric activity
Movement Sensors | 48 hours, 7 days, and 3 months poststroke
  Upper limb range of motion patterns
National Institutes of Health Stroke Scale | 48 hours, 7 days, and 3 months poststroke
  Neurological functions
Trunk Control Test | 48 hours, 7 days, and 3 months poststroke
  Sitting balance
Functional Ambulation Categories | 48 hours, 7 days, and 3 months poststroke
  Walking ability (independence)
Modified Rankin Scale | 48 hours, 7 days, and 3 months poststroke
  Global disability
Motor Activity Log - 14 | 48 hours, 7 days, and 3 months poststroke
  Patient-reported daily life upper limb use
Global Rating of Perceived Changes | 3 months poststroke
Concomitant Movement Therapy | 48 hours, 7 days, and 3 months poststroke
  Intensity of therapy based on charts
Safety | 48 hours, 7 days, and 3 months poststroke
  Serious Events (1. death; 2. life-threatening illness or injury; 3. in-patient or prolonged hospitalisation; 4. medical or surgical intervention to prevent life threatening illness; 5. led to fetal distress, death or a congenital abnormality or birth defect)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fattore G, Torbica A, Susi A, Giovanni A, Benelli G, Gozzo M, Toso V. The social and economic burden of stroke survivors in Italy: a prospective, incidence-based, multi-centre cost of illness study. BMC Neurol. 2012 Nov 14;12:137. doi: 10.1186/1471-2377-12-137. PMID 23150894
- [Background] Nijland RH, van Wegen EE, Harmeling-van der Wel BC, Kwakkel G; EPOS Investigators. Presence of finger extension and shoulder abduction within 72 hours after stroke predicts functional recovery: early prediction of functional outcome after stroke: the EPOS cohort study. Stroke. 2010 Apr;41(4):745-50. doi: 10.1161/STROKEAHA.109.572065. Epub 2010 Feb 18. PMID 20167916
- [Background] Stinear CM, Barber PA, Petoe M, Anwar S, Byblow WD. The PREP algorithm predicts potential for upper limb recovery after stroke. Brain. 2012 Aug;135(Pt 8):2527-35. doi: 10.1093/brain/aws146. Epub 2012 Jun 10. PMID 22689909
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539